CLINICAL TRIAL: NCT05520515
Title: Water and Land-based Aerobic Training on Health-related Outcomes in Breast Cancer Survivors: a Randomized Clinical Trial
Brief Title: Water and Land-based Aerobic Training in Breast Cancer Survivors
Acronym: WaterMama
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Cristine Lima Alberton, Principal Investigator, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 55791222.0.0000.5313
Record Dates: First submitted 2022-08-23; First posted 2022-08-30 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
Keywords: physical exercise; breast neoplasm; physical activity; aquatic exercise
MeSH Terms: conditions — Breast Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: The WaterMama trial is a randomized, single-blinded, three-arm, parallel, superiority trial. Forty-eight women, ≥18 years of age, who have completed primary treatment and been diagnosed with stage I-III breast cancer are recruited. Participants are randomly allocated on a 1:1:1 ratio to 12-week interventions of aerobic exercise training programs either on the aquatic or land environment two times per week plus health education, or an active-control group receiving health education intervention, once a week.
Who Masked: Outcomes Assessor
Masking Description: Blinding will be implemented for the outcome assessors. All tests and questionnaires will be supervised by an evaluator blinded to the participant's group. Due to the type of intervention, the investigator conducting exercise sessions and participants will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aquatic training plus health education group (Experimental): Aerobic exercise training program in the aquatic environment twice a week plus health education program once a week
  Interventions: Other: Aquatic Training Plus Health Education
- Land training plus health education group (Experimental): Aerobic exercise training program in the land environment twice a week plus health education program once a week
  Interventions: Other: Land Training Plus Health Education
- Health education group (Active Comparator): Health education program once a week
  Interventions: Other: Health Education

INTERVENTIONS:
Other: Aquatic Training Plus Health Education — Participants perform a 12-week training program with two weekly exercise sessions on non-consecutive days. Sessions last 45 min (5 min of warm-up, 35 min of exercise, and 5 min of stretching) throughout the intervention period. The intervention is performed at the thermal pool sector of Clube Brilhante in Pelotas city. The pool water temperature is maintained between 30-32°C, with participants immersed in the depth level between the xiphoid process and shoulders. The aquatic training group performs the following water aerobics exercises: stationary running, frontal kick, cross-country skiing, and butt kick during the stimulus and jumping jacks during the active recovery. The training session is collective, with 3 to 6 participants, supervised by two experienced instructors, one outside and one inside the pool. The group also receives the booklet and the offer of weekly meetings of an educational program (30 min before one of the training sessions) with the same interactive lectures.
  Arms: Aquatic training plus health education group
Other: Land Training Plus Health Education — Participants perform a 12-week training program with two weekly exercise sessions on non-consecutive days. Sessions last 45 min (5 min of warm-up, 35 min of exercise, and 5 min of stretching) throughout the intervention period. The intervention occurs at the School of Physical Education, Federal University of Pelotas. Depending on weather conditions, the land training group will perform aerobic training with walking/running exercises in a flat outdoor environment or inside a multi-sport gym. The training session will be collective, with 3 to 6 participants, supervised by two experienced instructors, one at the starting point and the other following the movement of the participants. In addition, the group receives the booklet and the offer of weekly meetings of an educational program (30 min before one of the training sessions) with the same interactive lectures.
  Arms: Land training plus health education group
Other: Health Education — The intervention occurs at the School of Physical Education, Federal University of Pelotas. The intervention consists of an educational program with weekly lectures of approximately 30 min. The lectures are led by a qualified health professional, using expository and interactive approaches on topics that cover basic knowledge related to breast cancer and complementary therapies. Additionally, each participant receives a self-care booklet containing information about the topics addressed during the meetings. Qualified professionals give lectures on the following topics: 1) fatigue and quality of life; 2) anxiety and depressive symptoms; 3) body image and sexual function; 4) self-esteem; 5) self-care; 6) sleep; 7) cognitive function; 8) symptoms in the arm and breast; 9) pain and arthralgia; 10) body composition and bone health; 11) eating habits; 12) physical activity.
  Arms: Health education group

SUMMARY:
Background: Breast cancer is the type of cancer that mostly affects women in the world. Although physical and psychological side effects accompany cancer and the aggressiveness of the treatment, regular practice of physical exercise is considered a non-pharmacological tool to improve the quality of life of breast cancer survivors. The present study aims to evaluate the effects of aerobic training programs in aquatic and land environments plus a health education program, compared with a health education program alone, on cancer-related fatigue and other health-related outcomes in breast cancer survivors.

Methods: The WaterMama trial is a randomized, single-blinded, three-arm, parallel, superiority trial. Forty-eight women, ≥18 years of age, who have completed primary treatment and been diagnosed with stage I-III breast cancer are recruited. Participants are randomly allocated on a 1:1:1 ratio to 12-week interventions of aerobic exercise training programs either on the aquatic or land environment two times per week plus health education, or an active-control group receiving health education intervention, once a week. Cancer-related fatigue (primary outcome), physical fitness (i.e., muscle strength of the knee extensors, muscle thickness and muscle quality of quadriceps, resting heart rate, maximum oxygen consumption, and performance in functional tests), mental health (i.e., depressive and anxiety symptoms), cognitive function, pain and quality of life are measured before and after 12 weeks of intervention. The analysis plan will use an intention-to-treat approach and protocol criteria.

Discussion: The conceptual hypothesis is that both training programs plus health education positively affect cancer-related fatigue, physical fitness, mental health, cognitive function, pain, and quality of life compared to the health education group alone. Additionally, it is expected that the aquatic program plus health education to provide more significant effects on cancer-related fatigue and physical parameters due to its multi-component character, with a consequent greater positive impact on other investigated parameters in this group.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with stage I-III breast cancer;
* Aged ≥ 18 years old;
* Have completed primary treatment for breast cancer (including surgery, chemotherapy, and/or radiotherapy) for at least six months and at most 12 months before the start of the intervention, regardless to be or not on hormonal treatment;
* Willingness to participate in either intervention group, as well as not to have a fear of the aquatic environment.

Exclusion Criteria:

* Presence of serious orthopedic, cardiovascular, or cardiopulmonary conditions that limit physical exercise participation;
* Major psychiatric or cognitive disorders;
* Active metastatic or locoregional disease;
* Severe nausea, anorexia, or another condition that makes it impossible to participate in the exercise;
* Engagement in regular exercise for more than 75 min weekly.
* Or were otherwise not cleared by their oncologist.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-12-19 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Cancer-related fatigue | Baseline (week 0) to post-training (week 13)
  Cancer-related fatigue is measured with the Portuguese Piper Fatigue Scale (PFS) version. The Brazilian version of the PFS is a valid and reliable instrument for assessing fatigue in cancer patients in Brazil (Mota et al., 2009). The PFS consists of 22 numerical items assessing fatigue experienced by the patients (Piper et al., 1998), using a 0-10 numeric scale. The PFS measures four dimensions of subjective fatigue are: behavioral/severity, affective meaning, sensory, and cognitive/mood. The total fatigue score is calculated by adding the four subscale scores and dividing this sum by four.

SECONDARY OUTCOMES:
Cardiorespiratory fitness | Baseline (week 0) to post-training (week 13)
  First, the participants are kept seated at rest for 5 min in a calm environment to take heart rate (HR) measurements at rest using a heart rate monitor (H10, Polar, Finland). Peak oxygen consumption (VO2peak), oxygen uptake in the first ventilatory threshold (VO2VT1) and oxygen uptake in the second ventilatory threshold (VO2VT2) are determined from a maximal incremental treadmill test (KIKOS, São Paulo - São Paulo, Brazil). Warming up is carried out for 3 min with a gradual increase in speed until reaching 3 km.h-1, and then the test starts at 3 km.h-1 with sequential increments of 0.5 km.h-1 every minute, and a 1% increase in grade every 2 min until maximum effort. The test is finished when the participant can no longer to exercise at a given workload, indicating exhaustion. All tests are supervised by a trained exercise physiologist and a physician.
Maximal dynamic strength | Baseline (week 0) to post-training (week 13)
  The maximum dynamic muscle strength of knee extensors will be measured through the one-repetition maximal test (1RM) performed in an extension chair. The 1RM value is considered the greatest load that the participant could lift for one complete repetition (i.e., concentric and eccentric phase) following a predetermined cadence (i.e., approximately 2 s per phase) controlled by a digital app (Metronome). The 1RM of each participant is determined within five attempts, and at least 3 min of rest interval was given between trials. A new load was estimated using correction factors (Lombardi, 1989) for the subsequent trial when the participant could perform more than one complete repetition. The test is rescheduled if the value of 1RM is not determined between the five attempts. According to a previous study from our laboratory (Andrade et al. 2020), the range of motion is individualized for each participant and controlled by a range of motion custom-build device.
Dynamic muscular endurance | Baseline (week 0) to post-training (week 13)
  The same knee extension machine is used to assess dynamic muscular endurance. To do so, participants perform the maximal number of bilateral knee extension repetitions at 60% of their 1RM. The test cadence (2 s for each contraction phase) and range of motion are the same for the 1RM test. The post-intervention assessment is performed using the same absolute load employed at baseline (i.e., 60% of baseline 1RM).
Functional tests - Arm Curl Test | Baseline (week 0) to post-training (week 13)
  The Arm Curl test is performed to measure the strength of the upper limbs. Starting at full elbow extension and holding a 2 kg dumbbell in each hand, participants are instructed to perform the maximal number of elbow crunches over the full range of motion for 30 s. The test is performed with both upper limbs.
Functional tests - 30-s Chair Stand Test | Baseline (week 0) to post-training (week 13)
  The 30-s Chair-Stand test is performed to measure the strength of the lower limbs. Participants are instructed to sit and stand up from a chair 43 cm high from the seat, without the aid of the upper limbs, as many times as possible during 30 s.
Functional tests - 8-ft Up and Go Test | Baseline (week 0) to post-training (week 13)
  The 8-ft Up-and-Go test is performed to measure agility and dynamic balance. Participants are instructed to get up from the chair (43 cm), turn around a marker that will be 2.44m, and return to the starting position. The shortest time of two attempts will be considered as a result.
Functional tests - Chair Sit-and-Reach Test | Baseline (week 0) to post-training (week 13)
  The Chair Sit-and-Reach test is performed to measure the flexibility of the lower limbs. Participants sit on the front edge of a chair and extend one leg straight out in front of the hip, with foot flexed and heel resting on the floor (the other leg is bent, foot flat on the floor). The object is to reach as far forward as possible toward (or past) the toes. The investigator uses a ruler noting the cm left to reach the toe (negative score) or the cm that went past the toe (positive score).
Functional tests - Back Scratch Test | Baseline (week 0) to post-training (week 13)
  The Back Scratch test is performed to measure the flexibility of the upper limbs. Participants are instructed to try to touch the middle fingers of both hands together behind the back. The investigator uses a ruler noting the cm left to reach the middle fingers (negative score) or the cm that the middle fingers overlapped (positive score).
Functional tests - 6-min Walk Test | Baseline (week 0) to post-training (week 13)
  The 6-min Walk test is performed to measure aerobic fitness. The course proposed in the original test is 45.72 m rectangular. The course will be adapted for a straight line with 30 m length, demarcated with cones every 3 m. Participants are instructed to walk for 6-min in a flat 30m course, in which the total distance walked "as fast as possible" is assessed.
Muscle thickness | Baseline (week 0) to post-training (week 13)
  Transversal images of the four portions of the quadriceps femoris are obtained by B-mode ultrasonography with a 7.5 megahertz linear array probe. Images of the vastus lateralis (VL), rectus femoris (RF), and vastus intermedius (VI) muscles are obtained at the midpoint between the anterosuperior iliac spine and the upper edge of the patella, whereas the vastus medialis (VM) is assessed at 30% of the distance between the lateral condyle and the greater trochanter of the femur. All images will be analyzed using the ImageJ software (National Institutes of Health, USA, version 1.37). The muscle thickness will be assessed as the distance from each muscle's superior and inferior muscle aponeurosis. Overall quadriceps femoris muscle thickness will be calculated as the sum of each muscle thickness (i.e., RF + VL + VM + VI).
Muscle quality | Baseline (week 0) to post-training (week 13)
  Transversal images of the four portions of the quadriceps femoris are obtained by B-mode ultrasonography with a 7.5 megahertz linear array probe. Images of the VL, RF, and VI muscles are obtained at the midpoint between the anterosuperior iliac spine and the upper edge of the patella, whereas the VM is assessed at 30% of the distance between the lateral condyle and the greater trochanter of the femur. All images will be analyzed using the ImageJ software. Muscle quality will be determined by the echo intensity values, which will be calculated from gray-scale analysis using the standard histogram function in ImageJ. The echo intensity of the quadriceps femoris will be calculated as the mean of echo intensity values of the four individual quadriceps femoris muscles ((RF + VL + VM + VI)/4).
Depressive and anxiety symptoms is measured using the Hospital Anxiety and Depression Scale (HADS). | Baseline (week 0) to post-training (week 13)
  HADS was developed by Zigmond and Snaith (1983), with translation and validation for the Brazilian population (Botega et al., 1995). It is an instrument composed of 14 items, seven of which form the anxiety subscale and the other seven the depression subscale, allowing the assessment of symptoms in the previous week. Each HADS item has four response options ranging from 0 to 3, reaching a maximum of 21 points in each subscale.
Perceived cognitive function | Baseline (week 0) to post-training (week 13)
  Aspects of perceived cognitive function will be measured using the Functional Assessment of Cancer Therapy - Cognitive Function - Version 3 questionnaire (FACT-Cog-v3). This instrument was developed specifically for cancer patients, consisting of 37 items, organized into four sections: perceived cognitive impairments, comments from others, perceived cognitive abilities and impact on quality of life (Wagner et al., 2009). Each FACT-Cog-v3 item has five response options (not at all = 0; a little bit = 1; somewhat = 2; quite a bit = 3; very much = 4), and the higher the score mean a better perceived cognitive function. The recall period should only consider the past 7 days.
Objective cognitive function - Trail Making Test (TMT) | Baseline (week 0) to post-training (week 13)
  Aspects of objective cognitive function are measured by the Trail Making Test (TMT). The version validated for the Brazilian population of TMT (Carvalho & Caramelli, 2020) is used to assess domains such as attention, motor skills, processing speed and cognitive flexibility (Bowie & Harvey, 2006). In the first part of the instrument (TMT-A), participants will have to draw a line connecting the numbers from 1 to 25 in ascending order. Then, letters (A-L) will be added so that the participants trace a line again following a numerical (1-13) and alphabetical order, interleaved (TMT-B). Participants will be instructed to maintain pencil-to-paper contact during the test. A shorter runtime indicates better performance.
Objective cognitive function - Controlled Oral Word Association Test (COWAT) | Baseline (week 0) to post-training (week 13)
  Aspects of objective cognitive function are also measured by the Controlled Oral Word Association Test (COWAT). The COWAT is used to assess verbal fluency, working memory and inhibitory control (Ross et al., 2007). In this test the participants will have to speak as many words as possible that start with the letters "F", "A" and "S", within 1 minute for each letter. Proper names, repeated words and variations in gender, number and conjugation will not be considered. The greater number of words evoked in each test indicates better verbal fluency.
Pain is characterized by the short version of the Brief Pain Inventory (BPI-B). | Baseline (week 0) to post-training (week 13)
  BPI-B is validated in Brazilian cancer patients (Ferreira et al., 2011). This instrument is composed of nine multidimensional items that assess: pain intensity, pain interference in the patient's life, pain location and treatments for pain control and relief (Cleeland & Ryan, 1994). The answers (scales from 0 to 10) should correspond to the pain felt at the time of the questionnaire and in the last 24 hours. The scores will be calculated by the average of the total of items. The higher the score, the greater the severity of pain.
Quality of life is measured using the Functional Assessment of Cancer Therapy-Breast questionnaire (FACT-B). | Baseline (week 0) to post-training (week 13)
  The FACT-B is a 37-item instrument designed to measure five domains of quality of life in breast cancer patients: physical (seven items), social/family (seven items), emotional (six items), functional (seven items) well-being, as well as a breast-cancer subscale (ten items). The answers are presented on a 5-point Likert scale. Participants are instructed to select the number that best represents their answer for the last seven days. Online written permission was obtained to use this questionnaire in the study. Its Portuguese-translated version is a valid and reliable tool (Michels et al., 2012).

OTHER OUTCOMES:
Body mass | Baseline (week 0) to post-training (week 13)
  Body mass measurements are performed using a digital scale with a stadiometer (WELMY, Santa Bárbara d'Oeste - São Paulo, Brazil). Body mass is measured in kilograms.
Height | Baseline (week 0) to post-training (week 13)
  Height measurements are performed using a digital scale with a stadiometer (WELMY, Santa Bárbara d'Oeste - São Paulo, Brazil). Height is measured in meters.
Body mass index | Baseline (week 0) to post-training (week 13)
  The calculation of the body mass index (BMI) is performed using the equation: BMI = body mass (kg)/height² (m).
Waist and hip circumferences | Baseline (week 0) to post-training (week 13)
  Waist and hip circumferences are measured with a measuring tape placed around the navel height and the width of the participants' hips, respectively, to calculate the waist-hip ratio.
Physical activity levels | Baseline (week 0) to post-training (week 13)
  The self-reported physical activity level is measured before and after 12 weeks of intervention using the Godin-Shephard Leisure-Time Physical Activity Questionnaire (Godin & Shephard, 1985). The translated and validated Brazilian version of the Godin-Shepard questionnaire is used (São-João et al., 2013). Participants should report the number of times a week they perform vigorous, moderate, and light physical activities for more than 15 minutes. The weekly frequencies of intense, moderate, and light activities should be multiplied by nine, five, and three, respectively. The total weekly leisure activity is calculated in arbitrary units from the sum of the products of each component.
Food consumption | Baseline (week 0) to post-training (week 13)
  The "Food frequency Questionnaire as subsidy for programs of non-communicable chronic diseases prevention" is used to control changes in food consumption (Ribeiro and Cardoso, 2002). The instrument is applied at baseline to provide the frequency of food consumption in the month before the intervention beginning and post-intervention to provide this information during the last month of intervention.
Office Blood Pressure | Baseline (week 0) to post-training (week 13)
  Systolic and diastolic blood pressure measurements are taken at baseline and after 12 weeks of intervention. Participants are kept in a calm environment for 5 min, and then a researcher measures the subject's BP using calibrated and automated oscillometric devices (OMRON Healthcare Inc., Bannockburn, USA) according to hypertension guidelines (Malachias et al., 2016). Initially, measurements are performed in both arms of the participant. After three measurements, with an interval of 1 to 2 min, are taken in the arm with the highest initial value. The average of the three measurements is considered the subject's office BP.
Sociodemographic and clinical characteristics | Baseline (week 0)
  Sociodemographic, reproductive, menstrual characteristics, family history of breast cancer, use of oral contraceptives, hormone replacement therapy, smoking, alcohol consumption are collected through a questionnaire administered before the intervention. Data on tumor histological type, tumor staging, hormone receptor status, and human epidermal growth factor receptor type 2 (HER-2) expression are collected from medical records.
Follow-up questionnaire | Post-training (week 13)
  Each participant answers 14 questions about individual perception related to the intervention using a Likert scale of 7 points, in which "1" means "no totally agreement" and "7" means "totally agreement". The questionnaire will be applied post-intervention to evaluate important outcomes in cancer patients such as safety, fun, motivation, future, benefits for daily life, intervention partner influence, training-related exhaustion, satisfaction, self-confidence on physical performance, supervision preference, changes in lifestyle, including physical activity and eating habits, and main barriers to group participation.
Adherence assessments | Post-training (week 13)
  Adherence measures are taken into account attendance and compliance in interventions. Attendance is monitored through the session's frequency recording and is treated as the percent of intervention sessions experienced by a participant given the total number of scheduled sessions (24 sessions for exercise programs or 12 sessions for the health education program). Compliance is treated as the percentage of intervention sessions entirely performed without protocol deviations.

CONTACTS AND LOCATIONS:
Overall Officials: Cristine L Alberton, PhD, Principal Investigator — Federal University of Pelotas; Stephanie S Pinto, PhD, Study Director — Federal University of Pelotas
Locations (1):
- Escola Superior de Educação Física, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alberton CL, Andrade LS, Xavier BEB, Pinheiro VHG, Cuesta-Vargas AI, Pinto SS. Land- and water-based aerobic exercise program on health-related outcomes in breast cancer survivors (WaterMama): study protocol for a randomized clinical trial. Trials. 2024 Aug 13;25(1):536. doi: 10.1186/s13063-024-08389-y. PMID 39138559